CLINICAL TRIAL: NCT02168881
Title: Oral Misoprostol Versus Vaginal Dinoprostone For Induction Of Labour: A Randomized Controlled Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Marwan Elkady, Dr, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Misoprostol-2014
Record Dates: First submitted 2014-06-19; First posted 2014-06-20 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Labour Induction
Keywords: labour; induction; misoprostol; dinoprostone
MeSH Terms: interventions — Misoprostol; Dinoprostone

ARMS (2):
- misoprostol (Active Comparator): oral misoprostol in solution 25 microgram every 2 hours
  Interventions: Drug: Misoprostol
- dinoprostone (Active Comparator): 3 mgs dinoprostone vaginally every six hours
  Interventions: Drug: Dinoprostone

INTERVENTIONS:
Drug: Misoprostol
  Arms: misoprostol
Drug: Dinoprostone
  Arms: dinoprostone

SUMMARY:
This study is to compare between oral misoprostol in solution and vaginal dinoprostone in induction of labour in primiparous women with singleton pregnancy as regards efficiency and safety to both mother and fetus.

ELIGIBILITY:
Inclusion Criteria:

* Primigravida
* >37 wks

Exclusion Criteria:

* Scarred uterus
* Macrosomia

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 342 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
induction delivery time | 2 hourly

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams Maternity hospital, Cairo, Egypt

REFERENCES:
- [Derived] Kerr RS, Kumar N, Williams MJ, Cuthbert A, Aflaifel N, Haas DM, Weeks AD. Low-dose oral misoprostol for induction of labour. Cochrane Database Syst Rev. 2021 Jun 22;6(6):CD014484. doi: 10.1002/14651858.CD014484. PMID 34155622